CLINICAL TRIAL: NCT04297319
Title: The Use of Laser in the Treatment of Atrophic Vulvovaginitis and Its Consequent Improvement in Sexual Satisfaction
Brief Title: The Use of Laser in the Treatment of Atrophic Vulvovaginitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This protocol was cancelled due to the COVID pandemic restrictions in our country. It was imposible to complete the recruitment of patients to achive the study objectives.
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, CLAUDIA ESTER MARCHITELLI, Chief of the Gynecology department, Hospital Italiano de Buenos Aires
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5076
Record Dates: First submitted 2019-11-05; First posted 2020-03-05 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Lasers; Atrophy of Vagina; Atrophy Vulva

STUDY DESIGN:
Intervention Model Description: Double blind, randomized, control clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The patient and the outcomes assessor and principal investigator has not access to the randomization system
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 - Laser intervention (Experimental): Laser diiodo treatment, 3 procedures of 5-10 minutes at intervals of 4 weeks
  Interventions: Procedure: Laser diiodo
- 2 - Laser placebo (Placebo Comparator): Only the laser speculum is placed in the vagina but the laser is not activated. 3 procedures of 5-10 minutes at intervals of 4 weeks
  Interventions: Procedure: Laser Placebo

INTERVENTIONS:
Procedure: Laser diiodo — 3 laser diiodo procedures of 5-10 minutes at intervals of 4 weeks It is an outpatient procedure, not anesthesia required.
  Arms: 1 - Laser intervention
Procedure: Laser Placebo — 3 laser diiodo procedures of 5-10 minutes at intervals of 4 weeks. It is an outpatient procedure, not anesthesia required.
  Arms: 2 - Laser placebo

SUMMARY:
This study evaluates the efficacy and security of laser for atrophy treatment. Half of participants will receive the laser treatment and the other half placebo.

DETAILED DESCRIPTION:
Thermal laser treatments are proposed as the newest treatments for atrophy. Through the thermal effect it would stimulates de mucosa, enhances the collagen component and the vascularization. Collagen remodeling and new collagen synthesis has been suggested as a mechanism of laser induced skin resurfacing and remodeling of vaginal connective tissue.

ELIGIBILITY:
Inclusion Criteria:

* Menopause women with vulvovaginal symptoms of atrophy
* No previous estrogen treatment for the last 30 days
* Active sexual life (vaginal penetration)
* Accept to participate
* Pap atrophy or hypotrophy in the last year

Exclusion Criteria:

* Vulvovaginal diseases
* Abnormal uterine bleeding
* Antidepressants drugs
* Uncontrolled diabetes
* Cervical intraepithelial lesions or cancer
* Photosensitized or under treatment with photosensibilized drugs
* Collagen diseases
* Vulvovaginal infections in the last 15 days
* Immunosuppressed patients or under immunosuppressed treatments

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Female Sexual Function Index questionnaire | baseline, and week 4 after treatment
  Female Sexual Function Index is a self- administered questionnaire that evaluate 19 items about sexual life. Minimum score is 2, and the highest is 36. Higher score mean a better outcome
Change from Baseline in Female Sexual Function Index questionnaire | baseline,and week 12 after treatment
  Female Sexual Function Index is a self- administered questionnaire that evaluate 19 items about sexual life. Minimum score is 2, and the highest is 36. Higher score mean a better outcome
Change from Baseline in Female Sexual Function Index questionnaire | baseline, and week 36 after treatment
  Female Sexual Function Index is a self- administered questionnaire that evaluate 19 items about sexual life. Minimum score is 2, and the highest is 36. Higher score mean a better outcome
Vaginal Cytology Improvement | baseline, and week 4 after treatment
  Vagina cytology will be obtain to evaluate initial conditions of the vagina and modifications after treatment. Papanicolaou coloration and the count of superficial, intermediate, parabasal and basal cells will be applied to measure improvement of vaginal atrophy
Vaginal Cytology Improvement | baseline, and week 12 after treatment
  Vagina cytology will be obtain to evaluate initial conditions of the vagina and modifications after treatment. Papanicolaou coloration and the count of superficial, intermediate, parabasal and basal cells will be applied to measure improvement of vaginal atrophy
Vaginal Cytology Improvement | baseline, and week 36 after treatment
  Vagina cytology will be obtain to evaluate initial conditions of the vagina and modifications after treatment. Papanicolaou coloration and the count of superficial, intermediate, parabasal and basal cells will be applied to measure improvement of vaginal atrophy
Change in vaginal acidity measure | baseline, and week 4 after treatment
  the normal vaginal acidity is between 3,8 a 4,5. In postmenopausal women is higher. We are going to evaluate the improvement in vaginal acidity to normal values of premenopausal women. It will be evaluate with specific acidity measurement strips (this strips measures between 3.8 y 5.4)
Change in vaginal acidity measure | baseline, and week 12 after treatment
  the normal vaginal acidity is between 3,8 a 4,5. In postmenopausal women is higher. We are going to evaluate the improvement in vaginal acidity to normal values of premenopausal women. It will be evaluate with specific acidity measurement strips (this strips measures between 3.8 y 5.4)
Change in vaginal pH measure | baseline,and week 36 after treatment
  the normal vaginal ph is between 3,8 a 4,5. In postmenopausal women is higher. We are going to evaluate the improvement in vaginal acidity to normal values of premenopausal women. It will be evaluate with specific acidity measurement strips (this strips measures between 3.8 y 5.4)

SECONDARY OUTCOMES:
Number of patient with Local Estrogen therapy requirement post intervention | baseline,and week 48
  Number of patients that Need estrogen replacement for atrophy vulvovaginal symptoms, despite the intervention.This will be evaluate with a Yes/No question.

OTHER OUTCOMES:
Number of participant with Adverse events reported in each visit | Baseline,and week 48
  It will be evaluate the number of patients that reported adverse events such as dyspareunia, irritation, edema, vaginal dryness, genital bleeding, vaginal discharge, pain, lesions

CONTACTS AND LOCATIONS:
Overall Officials: claudia E Marchitelli, MD, Principal Investigator — Hospital Italiano de Buenos Aires, Argentina
Locations (1):
- Hospital Italiano de Buenos Aires, CABA, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Knight C, Logan V, Fenlon D. A systematic review of laser therapy for vulvovaginal atrophy/genitourinary syndrome of menopause in breast cancer survivors. Ecancermedicalscience. 2019 Dec 12;13:988. doi: 10.3332/ecancer.2019.988. eCollection 2019. PMID 32010212
- [Result] Adabi K, Golshahi F, Niroomansh S, Razzaghi Z, Ghaemi M. Effect of the Fractional CO2 Laser on the Quality of Life, General Health, and Genitourinary Symptoms in Postmenopausal Women With Vaginal Atrophy: A Prospective Cohort. J Lasers Med Sci. 2020 Winter;11(1):65-69. doi: 10.15171/jlms.2020.11. Epub 2020 Jan 18. PMID 32099629